CLINICAL TRIAL: NCT05751291
Title: Comparative Study to Evaluate the Efficacy of Ultrasound-Guided Pericapsular Nerve Group (PENG) Block Versus Fascia Iliaca Compartment (FIC) Block on the Postoperative Analgesic Effect in Patients Undergoing Hip Surgeries Under Spinal Anesthesia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Kamed Mohamed, Comparative Study to Evaluate the Efficacy of Ultrasound-Guided Pericapsular Nerve Group (PENG) Block Versus Fascia Iliaca Compartment (FIC) Block on the Postoperative Analgesic Effect in Patients Undergoing Hip Surgeries under Spinal Anesthesia., Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-02-08
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A (PENG block) patients will receive PENG block under ultrasound-guided (USG) guidance using curvilinear low-frequency ultrasound probe (2-5 MHz) will initially be placed in a transverse plane over the Anterior inferior iliac spine ( AIIS ) and then aligned with the pubic ramus by rotating the probe counterclockwise approximately 45 degrees to visualize the Iliopubic Eminence (IPE), the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle. A 22 Gauge needle will be inserted in-plane and the needle tip will be positioned in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. 20 mL of 0.25% bupivacaine will be injected in increments while observing for an adequate fluid spread in this plane.
  Interventions: Drug: Bupivacaine Hydrochloride
- Group B (Active Comparator): Group B (FIC) patients will receive FIC block under USG guidance using high-frequency linear transducer (6-13 MHz) will be used to identify the femoral artery at the level of the inguinal crease. Immediately lateral and deep to the femoral artery and vein the iliopsoas muscle is overlaid by a hyperechoic fascia iliaca. The femoral nerve is seen lateral to the femoral artery wedged between the iliopsoas muscle and the fascia iliaca.
  Maneuvering the transducer laterally helps to visualize the Sartorius muscle covered by its own fascia alongside the fascia iliaca. A line is drawn connecting the anterior superior iliac spine to the pubic tubercle; the needle tip is positioned at lateral third of the line under the fascia iliaca. 20 mL of 0.25% bupivacaine will be injected until it spreads laterally toward the iliac spine and medially toward the femoral nerve.
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — Pericapsular Nerve Group (PENG) Block: 20 mL of 0.25% bupivacaine will be injected in increments while observing for an adequate fluid spread in this plane. Fascia Iliaca Compartment (FIC) Block: 20 mL of 0.25% bupivacaine will be injected until it spreads.
  laterally toward the iliac spine and medially toward the femoral nerve.

SUMMARY:
Fractures in and around the hip are quite common irrespective of both the young and elderly population groups and are associated with extreme pain. A hip fracture is a serious injury, with complications that can be life-threatening and is a common orthopedic emergency in the elderly. Early surgery within 48 h of fracture has shown to decrease the complication and mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* Forty -Two patients above 18 years of age belonging to the American Society of Anaesthesiologists (ASA) physical status Classes I and II scheduled for hip surgery will randomly be allocated into two groups. Group A (PENG block) will receive US - guided PENG block and Group B (FIC block) will receive US - guided FIC block for postoperative pain relief.

Exclusion Criteria:

* Patient refusal.
* Patient with significant neurological, psychiatric or neuromuscular disease.
* Alcoholism.
* Drug abuse.
* Pregnancy or lactating women.
* Suspected Coagulopathy.
* Morbid obesity.
* Known allergy to study medications.
* Septicemia and local infection at the block site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between duration of analgesia of Pericapsular Nerve Group (PENG) Block vs Fascia Iliaca Compartment (FIC) Block. | 6 months
  Comparison between duration of analgesia of Pericapsular Nerve Group (PENG) Block vs Fascia Iliaca Compartment (FIC) Block.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] WERTHEIMER LG. The sensory nerves of the hip joint. J Bone Joint Surg Am. 1952 Apr;34-A(2):477-87. No abstract available. PMID 14917714
- [Background] GARDNER E. The innervation of the hip joint. Anat Rec. 1948 Jul;101(3):353-71. doi: 10.1002/ar.1091010309. No abstract available. PMID 18873153
- [Background] Gerhardt M, Johnson K, Atkinson R, Snow B, Shaw C, Brown A, Vangsness CT Jr. Characterisation and classification of the neural anatomy in the human hip joint. Hip Int. 2012 Jan-Feb;22(1):75-81. doi: 10.5301/HIP.2012.9042. PMID 22344482
- [Background] Short AJ, Barnett JJG, Gofeld M, Baig E, Lam K, Agur AMR, Peng PWH. Anatomic Study of Innervation of the Anterior Hip Capsule: Implication for Image-Guided Intervention. Reg Anesth Pain Med. 2018 Feb;43(2):186-192. doi: 10.1097/AAP.0000000000000701. PMID 29140962